CLINICAL TRIAL: NCT06752408
Title: Aumolertinib Versus Osimertinib As First-line Therapy for Patients with EGFR Mutated Locally Advanced or Metastatic Non-small-cell Lung Cancer: a Randomized, Open-label, Non-inferiority Real World Study
Brief Title: Aumolertinib Versus Osimertinib As First-line Therapy for Patients with EGFR Mutated Locally Advanced or Metastatic Non-small-cell Lung Cancer
Acronym: ANOTHER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University People's Hospital (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wang mengzhao, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K6674
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; EGFR mutation; Aumolertinib; Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aumolertinib (Experimental)
  Interventions: Drug: Aumolertinib
- Osimertinib (Active Comparator)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Aumolertinib — Aumolertinib will be administered orally at a dose of 110 mg per time, Q.D.
  Arms: Aumolertinib
Drug: Osimertinib — Osimertinib will be administered orally at a dose of 80 mg per time, Q.D.
  Arms: Osimertinib

SUMMARY:
This is a multicenter, randomized, open-label, non-inferiority real world study. The study is designed to evaluate the efficacy and safety of Aumolertinib versus Osimertinib in the first-line treatment of patients with EGFR mutated locally advanced or metastatic non-small-cell lung cancer.

DETAILED DESCRIPTION:
Aumolertinib and Osimertinib are both third-generation, irreversible epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) that were approved for non-small cell lung cancer (NSCLC) patients with EGFR mutation.

This study will compare the efficacy of two different EGFR-TKIs, Aumolertinib and Osimertinib, when administered as monotherapy.

This is a multicenter, randomized, open-label study with 2 different groups that are listed below.

In a randomized study, the treatment that participants receive is randomly assigned, with the assignment determined by a computer algorithm. In an "open-label" study, both the participants and the investigators are aware of the treatment allocation for each participant.

Participants will be randomly assigned to one of the following two treatment groups:

Group 1: Treatment with Aumolertinib alone, taken orally as two pills once a day. Around 158 participants will be randomly assigned to this group.

Group 2: Treatment with Osimertinib alone, taken orally as one pill once a day. Around 158 participants will be randomly assigned to this group.

Participants can continue to receive treatment as long as they have not withdrawn consent, as long as they choose to continue to receive treatment and are judged by their doctor to continue to receive clinical benefit from receiving the treatment, and as long as no other exclusion and/or discontinuation criteria are met .

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Participants voluntarily signed an informed consent form prior to participation.
3. The Eastern Cooperative Oncology Group (ECOG) physical status score of 0 or 1, no deterioration for at least 1 week before treatment, and the expected survival period is no less than 12 weeks.
4. Histologically or cytologically confirmed stage IIIB-IV NSCLC (according to the AJCC eighth edition lung cancer staging criteria), metastatic or recurrent lung cancer that is not amenable to curative intent therapy.
5. Positive EGFR mutation confirmed by tissue or cytology(including peripheral blood, pleural effusion, ascites, cerebrospinal fluid) with at least one sensitizing mutation (L858R or 19Del).
6. No prior systemic therapy was allowed, except in the adjuvant or neoadjuvant setting, and no progression was allowed within 6 months.
7. According to RECIST1.1, the patient must have at least one target lung lesion. The requirements for target lesions are: measurable lesions that have not undergone local treatment such as radiation, with the longest diameter at baseline ≥10 mm (if it is a lymph node, the maximum short diameter must be ≥15 mm).

Exclusion Criteria:

1. Diagnosis of meningeal metastasis by clinical symptoms or imaging or cerebrospinal fl-uid, or brain parenchymal metastasis combined with meningeal metastasis.
2. History of other primary malignant tumors.
3. Hypersensitivity or allergy to aumolertinib or osimertinib or their excipients.
4. Female subjects who are pregnant, lactating, or planning to become pregnant during the treatment period.
5. The investigator assesses whether there are any patients with conditions that may compromise patient safety or interfere with the evaluation of the study, such as poorly controlled hypertension, active bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-12-17 (Estimated); Primary Completion 2027-01-16 (Estimated); Study Completion 2028-01-16 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Investigator Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 3 years
  PFS is defined as the time from date of randomization until date of disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from date of randomization until death from any cause.
Objective Response Rate (ORR) as Assessed by Investigator Per RECIST v1.1 | Up to 3 years
  ORR is defined as proportion of participants who achieve a complete response or partial response at any time before progressive disease or initiating a subsequent anticancer therapy.
Disease Control Rate (DCR) as Assessed by Investigator Per RECIST v1.1 | Up to 3 years
  DCR is defined as the proportion of participants who have a best overall response of complete response or partial response or stable disease.
Duration of Response (DOR) as Assessed by Investigator Per RECIST v1.1 | Up to 3 years
  DOR is defined as date of first response (complete response or partial response) until date of disease progression or death due to any cause, whichever occurs first.
Depth of Response (DepOR) as Assessed by Investigator Per RECIST v1.1 | Up to 3 years
  DepOR is defined as the relative change in target lesion tumor size (calculated as the sum of the longest diameters of the target lesions, in the absence of new lesions or progression of nontarget lesions) as compared to baseline.
Treatment-emergent adverse events (TEAEs) | From first dose until 28 days after the last dose, up to 36 month
  This outcome measures the type, incidence, grade and severity of treatment-emergent adverse events (TEAEs) that occur during treatment (as determined by the NCI-CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Undecided